CLINICAL TRIAL: NCT00557713
Title: Treatment of Induction With XELOX-Bevacizumab in Locally Advanced Rectal Adenocarcinoma: Phase II Study
Brief Title: XELOX+Bevacizumab Followed by Capecitabine+Bevacizumab+Radiotherapy as Neoadjuvant Treatment of Locally Advanced Rectal Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associacio catalana per a la recerca oncologica i les seves implicacions sanitaries i socials (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVACROSS
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Rectal Neoplasms; Locally Advanced Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): 1. -Induction treatment. 4 cycles (every 3 weeks) of bevacizumab (7,5mg/kg day 1) + oxaliplatin (130mg/m2 day 1) + capecitabine (1000mg/m2/12h days 1-14)
  2. -Concomitant (CT+RT) treatment (3 weeks later): bevacizumab (5mg/kg day 1 of 1st, 3th and 5th weeks) + capecitabine (825mg/m2/12h daily during radiotherapy treatment) + radiotherapy (45Gy (25fractions of 1,8Gy/day over 5weeks) followed by boost 5.4Gy (1,8Gy/day over 3days))
  3. -Surgery (6-8 weeks after last bevacizumab dose)
  4. -Adjuvant treatment: It will be individual decision of each investigator, but it's recommended 4 cycles of XELOX (equal dose at induction treatment)
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — 1. -Induction treatment. 4 cycles (every 3 weeks) of bevacizumab (7,5mg/kg day 1) + oxaliplatin (130mg/m2 day 1) + capecitabine (1000mg/m2/12h days 1-14)
  2. -Concomitant (CT+RT) treatment (3 weeks later): bevacizumab (5mg/kg day 1 of 1st, 3th and 5th weeks) + capecitabine (825mg/m2/12h daily during radiotherapy treatment) + radiotherapy (45Gy (25fractions of 1,8Gy/day over 5weeks) followed by boost 5.4Gy (1,8Gy/day over 3days))
  3. -Surgery (6-8 weeks after last bevacizumab dose)
  4. -Adjuvant treatment: It will be individual decision of each investigator, but it's recommended 4 cycles of XELOX (equal dose at induction treatment)
  Other Names: Avastin

SUMMARY:
The purpose of this study is to determine the pathological complete response rate of addition of bevacizumab to induction therapy (xelox) and concomitant treatment (capecitabine+radiotherapy), followed by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from patients who are able to understand the study request
* Histologically confirmed diagnosis of locally advanced rectal adenocarcinoma; ≤12 cm from the anal margin; T3, operable T4 or TxN+
* Karnofsky PS Index ≥ 70%
* Life expectancy > 6 months
* Adequate bone marrow, liver and renal function: ANC ≥ 1.5 x 10e9/l; Platelets ≥ 100 x 10e9/l; Hb ≥ 9g/dl; INR ≤ 1.5; Bilirubin ≤ 1.5 x ULN; ALT and/or AST ≤ 2.5 x ULN or ≤ 5 x ULN (in case of hepatic metastasis); Alkaline phosphatase ≤ 2.5 x ULN or ≤ 5 x ULN (in case of hepatic metastasis) or ≤ 10 x ULN (in case of bone metastasis); Creatinine clearance (Cockcroft-Gault) ≥ 30 ml/min or seric creatinine ≤ 1.5 x ULN

Exclusion Criteria:

* Distant metastases; previous neoplasm during last 5 years or previous infiltrating neoplasm; previous treatment with radiotherapy or study drugs; recruited for other clinical trial in 4 weeks before study entry
* Surgery, open biopsy or traumatic injury in 4 weeks before study entry; fine-needle aspiration in 7 days before study entry; major surgery planned during study
* Previous heart disease or uncontrolled hypertension, previous hemorrhagic diathesis or coagulopathy; full-dose oral or parenteral anticoagulant or thrombolytic agent (low-dose warfarin is allowed, INR ≤ 1.5); chronic use of high-dose aspirin (<325mg/day) or non-steroidal anti-inflammatory treatment
* No integrity of the upper gastrointestinal tract, malabsorption syndrome or unable to take oral drugs
* Pregnant or lactating patients; SNC disease; allogeneic transplant with immunosuppressive drugs; bone fracture not healed, wound or severe ulcers; uncontrolled intercurrent severe infections; previous related-fluoropyrimide SAEs or DPD deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2007-02; Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | after concomitant CT-RT treatment

SECONDARY OUTCOMES:
Complete Resection (R0) Rate | after surgery
Disease Free Survival | from complete response to relapse or disease-related death
Time to Failure Treatment | from first treatment dose to drop out of the study
Metastatic or Local Recurrence | during study
Toxicity Evaluation | during study
Surgical Morbility | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Nogué, MD, Study Chair — Associacio catalana per a la recerca oncologica i les seves implicacions sanitaries i socials
Locations (1):
- ACROSS, Barcelona, Spain

REFERENCES:
- See also: across — http://www.acrosscancer.org